CLINICAL TRIAL: NCT02329756
Title: Tranexamic Acid in Adherent Placenta (TAP), a Randomized Clinical Trial
Brief Title: Tranexamic Acid in Adherent Placenta (TAP)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: More preparation needed prior to collecting data.
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Karin Anneliese Fox M.D., M.Ed., Assistant Professor Obstetrics and Gynecology, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-41847; H-41847 (Other: Baylor College of Medicine Institutional Review Board)
Record Dates: First submitted 2014-12-29; First posted 2015-01-01 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Placenta Accreta
Keywords: Tranexamic Acid
MeSH Terms: conditions — Placenta Accreta | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study drug and placebo will be prepared by Investigational Pharmacy, and with similar appearing packaging and syringes. The Investigational Pharmacy will maintain the randomization table and allocation list. Participants, care providers, investigators and outcomes assessors will remain blinded until after data analysis completed, unless unblinding required in case of clinical emergency, per the unblinding procedures within the protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment (Active Comparator): Tranexamic acid (TXA) will be compared with matching placebo (sodium chloride 0.9%).
  Interventions: Drug: Tranexamic Acid (TXA)
- Control (Placebo Comparator): Matching placebo (sodium chloride 0.9%) will be compared with treatment group
  Interventions: Drug: Sodium Chloride 0.9%

INTERVENTIONS:
Drug: Tranexamic Acid (TXA) — 1g Tranexamic Acid (TXA) will be given at the time of delivery. If in 30 minutes, heavy bleeding continues, a 2nd dose will be administered.
  Other Names: Cyklokapron
  Arms: Treatment
Drug: Sodium Chloride 0.9% — Dose 1: 1 gram - to be administered by intravenous injection at an approximate rate of 1 mL/minute to all randomized women approximately 10 minutes prior to induction of anesthesia
  Dose 2: 1 gram - If 30 minutes after beginning the cesarean section there is significant bleeding as defined by the need for the transfusion of 4 or more units of blood products, or if there is a rebleed within the 24 hours after the first dose, a second dose may be given. To be administered by intravenous injection at an approximate rate of 1 mL/minute.
  The trial treatment injections should not be mixed with blood for transfusion, or infusion solutions containing penicillin or mannitol.
  Other Names: NaCl
  Arms: Control

SUMMARY:
The objective of this study is to investigate the effect of tranexamic acid (TXA) administration on the outcome of cesarean-hysterectomy in women with suspected Morbidly Adherent Placenta (MAP; placenta accreta, increta, percreta).

DETAILED DESCRIPTION:
This trial is a randomized, double blind, placebo controlled trial to quantify the effects of the preoperative administration of tranexamic acid on estimated blood loss and blood product utilization in women undergoing cesarean-hysterectomy for suspected MAP. Subgroup analyses will be performed for laboratory results (coagulation studies, electrolytes, complete blood count), urine output, hemodynamic parameters, return to OR for continued bleeding, post-operative complications (thromboembolism, wound separation, infection, fever), and length of hospital stay. Eligible patients will be randomized to receive either TXA or placebo.

Women eligible for inclusion will be identified during their prenatal course or on admission to the hospital prior to surgery. They will be offered participation in the study after appropriate counseling regarding the equipoise regarding TXA and its use in pregnancy, and following a question and answer period they will be consented, and assigned a study number.

A randomization table will be generated by the Texas Children's Hospital Investigational Pharmacy, using balanced blocks of 8, and will maintain control of the randomization to ensure blinding of participants and the clinical investigators. Randomization will occur when an order for study medication will be sent on a paper requisition to the Texas Children's Hospital Investigational Pharmacy, and a randomization number will be assigned to correspond to the study number. Ideally, this order will be sumbitted 24h prior to scheduled surgery, but may be submitted for urgent cases by calling the Texas Children's Clinical Pharmacy, and delivering the paper requisition to the 7th Floor Main Pharmacy.

The Investigational Pharmacy will prepare study medication (Tranexamic acid I.V. or Normal saline as placebo) as determined by the randomization. The medication (whether study medication or placebo) will be packaged in identical syringes. Sealed, opaque envelopes will be available to the PI or an assigned designee to permit unblinding (linking randomization number and study number) only in the event of a clinical emergency involving a study partipant during times at which the Investigational Pharmacy is closed (nights, weekends, holidays).

Once a patient has been randomized, the outcome in hospital will be collected even if the study medication is interrupted or not actually given.

ELIGIBILITY:
Inclusion Criteria:

* Ultrasound and/or MRI diagnosed MAPL pregnancy scheduled to have a cesarean hysterectomy
* The responsible clinician is substantially uncertain as to whether or not to use TXA
* Consent has been given according to approved procedures

Exclusion Criteria:

* Women for whom the responsible clinician considers there is a clear indication for TXA should not be randomized
* Prior known thromboembolic event during pregnancy
* Known contraindication to TXA (prior adverse reaction)
* Patient unable to give adequate consent due to emergent cesarean hysterectomy
* Bleeding prior to incision
* Prior known thromboembolic event
* Women with a history of any acute venous or arterial thrombosis including retinal artery/retinal vein occlusion, cerebrovascular accident, myocardial infarction, deep venous thrombosis, pulmonary embolism
* History of decreased renal function, renal cortical disease, or significant renal tract disease.

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The inclusion criteria includes pregnant women.
Enrollment: 0 (Actual)
Dates: Start 2018-12 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Estimated blood loss (EBL) | At patient discharge, upon death or 6 weeks (42 days) after randomization, whichever occurs first
  Our data from the past 65 cases of MAPL performed by our team over the past 3 years shows a 2500 +/- 500ml mean blood loss with these surgeries. Using pooled estimates of the reduction in blood loss published in the literature, a 30% reduction is a reasonable expectation.
Blood product requirements | At patient discharge, upon death or 6 weeks (42 days) after randomization, whichever occurs first
  The administration of a fixed dose is more practicable in this study and we have thus selected a fixed dose of 1 gram of TXA 10 minutes prior to induction of anesthesia, followed by a second dose of 1 gram if heavy bleeding is encountered 30 or more minutes after starting the cesarean section which requires the transfusion of 4 or more units of blood products. This is within the dose range which has been shown to inhibit fibrinolysis and provide hemostatic benefit.
Hemoglobin level change post surgery | At patient discharge, upon death or 6 weeks (42 days) after randomization, whichever occurs first
  The level of hemoglobin change will be measured after surgery.

SECONDARY OUTCOMES:
Thromboembolic events | From time patient is given treatment up to 12 weeks post-partum.
  Data from all thromboembolic events will be documented on CRFs, including but not limited to the amount and severity of events.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Belfort, MD, PhD, Principal Investigator — Baylor College of Medicine; Karin A Fox, MD,MEd, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No